CLINICAL TRIAL: NCT03267511
Title: A Randomized, Examiner-blind, Proof of Principal Study to Investigate the Stain and Plaque Removal Capability of Two Experimental 5% Potassium Nitrate Dentifrices in Healthy Subjects With the Propensity for Extrinsic Dental Stain
Brief Title: A Study to Investigate the Stain and Plaque Removal Capability of Two Experimental Potassium Nitrate Dentifrices
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 208078
Record Dates: First submitted 2017-08-28; First posted 2017-08-30 (Actual); Results first posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Oral Hygiene

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Test Product 1 (Experimental): Participants will be instructed to apply experimental dentifrice containing 5% potassium nitrate (KNO3) / 0.2542% sodium fluoride (NaF) dentifrice with 0.5% spherical silica.
  Interventions: Drug: 5% KNO3 / 0.2542% NaF dentifrice with 0.5% spherical silica
- Test Product 2 (Experimental): Participants will be instructed to apply experimental dentifrice containing 5% KNO3 / 0.2542% NaF dentifrice with 1% spherical silica and 5% STP.
  Interventions: Drug: 5% KNO3 / 0.2542% NaF dentifrice with 1% spherical silica and 5% STP
- Reference Product 1 (Active Comparator): Participants will be instructed to apply experimental dentifrice containing 5% KNO3 / 0.2542% NaF dentifrice with 6% abrasive silica.
  Interventions: Drug: 5% KNO3 / 0.2542% NaF dentifrice with 6% abrasive silica
- Reference Product 2 (Active Comparator): Participants will be instructed to apply experimental dentifrice containing 5% KNO3 / 0.2543% NaF dentifrice with 16% abrasive silica and 5% STP.
  Interventions: Drug: 5% KNO3 / 0.2543% NaF dentifrice with 16% abrasive silica and 5% STP

INTERVENTIONS:
Drug: 5% KNO3 / 0.2542% NaF dentifrice with 0.5% spherical silica — Participants will be instructed to apply a full brush head of their dentifrice containing 5% KNO3 / 0.2542% NaF dentifrice with 0.5% spherical silica and brush twice daily (morning and evening) for one timed minute (in their usual manner).
  Arms: Test Product 1
Drug: 5% KNO3 / 0.2542% NaF dentifrice with 1% spherical silica and 5% STP — Participants will be instructed to apply a full brush head of their dentifrice containing 5% KNO3 / 0.2542% NaF dentifrice with 1% spherical silica and 5% STP and brush twice daily (morning and evening) for one timed minute (in their usual manner).
  Arms: Test Product 2
Drug: 5% KNO3 / 0.2542% NaF dentifrice with 6% abrasive silica — Participants will be instructed to apply a full brush head of their dentifrice containing 5% KNO3 / 0.2542% NaF dentifrice with 6% abrasive silica and brush twice daily (morning and evening) for one timed minute (in their usual manner).
  Arms: Reference Product 1
Drug: 5% KNO3 / 0.2543% NaF dentifrice with 16% abrasive silica and 5% STP — Participants will be instructed to apply a full brush head of their dentifrice containing 5% KNO3 / 0.2543% NaF dentifrice with 16% abrasive silica and 5% STP and brush twice daily (morning and evening) for one timed minute (in their usual manner).
  Arms: Reference Product 2

SUMMARY:
The purpose of this study is to determine whether spherical silica can achieve similar or greater extrinsic dental stain and plaque removal, in comparison to dentifrices containing higher concentrations of standard abrasive silica, and how the addition of 5% sodium tripolyphosphate (STP) enhances cleaning capability.

DETAILED DESCRIPTION:
This proof of principal (PoP) single centre, randomised, examiner blind, four-treatment arm, parallel design study will be conducted in healthy participants with a propensity for extrinsic dental stain (based on the judgement of the examiner) on the facial surfaces of the anterior teeth. This study will be used to evaluate and compare the extrinsic dental stain and plaque removal of an experimental low abrasivity 0.5% spherical silica dentifrice and a marketed low abrasivity 6% standard silica abrasive dentifrice, and an experimental moderate abrasivity 1% spherical silica / 5% STP dentifrice and a marketed high abrasivity 16% standard abrasive silica / 5% STP dentifrice. Stain will be assessed using an established clinical measure of extrinsic dental stain - the MacPherson modification of the Lobene stain index (MLSI). Particpants will be stratified by baseline MLSI score (total MLSI (area [A] × intensity [I]) for the facial surfaces of the 4 anterior assessment teeth). Plaque will be assessed using an established clinical measure of plaque - the Turesky Modification of the Quigley Hein Index. Stain and plaque will be assessed at intervals over an 8 week treatment period. Plaque will be assessed at baseline and Week 8 only.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study before any assessment is performed.
* Male and female participants who, at the time of screening, are between the ages of 18 and 65 years, inclusive.
* Participants who are willing and able to comply with scheduled visits, treatment plan, and other study procedures.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee no clinically significant and relevant abnormalities of medical history or oral examination which could impact study outcomes.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee an absence of any condition that would impact on participant safety or wellbeing, or affect the participant's ability to understand and follow study procedures and requirements.
* In the opinion of the investigator or medically qualified designee, at screening, participants must have good oral health.
* In the opinion of the investigator or medically qualified designee, at screening, participants must have at least 20 natural teeth including the 12 anterior teeth, gradable for Turesky Plaque Index (TPI) (Gradable teeth are those where restorative materials cover less than 25% of the tooth surface to be graded).
* In the opinion of the investigator or medically qualified designee, at screening, participants must have the facial surfaces of at least 4 of the anterior teeth, gradable for the MLSI.
* In the opinion of the investigator or medically qualified designee, at screening, participants must have the presence of extrinsic dental stain (judged to be formed due to dietary factors) on the facial surfaces of the anterior teeth, as determined from a visual MLSI stain assessment.
* In the opinion of the investigator, at Visit 2, participants must have a sufficient level of extrinsic dental stain (in the opinion of the examiner) on the facial surfaces of the scorable anterior (maxillary and mandibular) teeth.
* At Visit 3, a minimum overall pre-brushing plaque score (TPI) of ≥2.0.

Exclusion Criteria:

* Participants who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or participants who are GSK employees directly involved in the conduct of the study.
* Participation in another clinical study or receipt of an investigational drug(s) within 30 days prior to study entry and/or during study participation.
* Participants who have previously been enrolled in this study.
* Acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Any condition which, in the opinion of the investigator, causes xerostomia.
* Pregnant female participants.
* Breastfeeding female participants.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Unwilling or unable to comply with the lifestyle guidelines described in this protocol.
* Recent history (within the last year) of alcohol or other substance abuse.
* Participant is unwilling to abstain from tobacco or nicotine-containing product use (including E-cigarettes) during the treatment evaluation period.
* Participants using the following mouth rinses, or taking the medications listed below: a) Regular use of mouthwashes containing ingredients that are known to impart staining. For example, chlorhexidine, essential oils or cetylpyridinium chloride (CPC). b) Use of a chlorhexidine, essential oil or CPC containing mouthwash within 14 days of Visit 2 or throughout the study. c) Current use of Listerine, or any antimicrobial mouth rinse. d) Use of minocycline, tetracycline or doxycycline within 30 days prior to screening. e) Use of minocycline, tetracycline or doxycycline between the screening and baseline visits. f) Daily doses of a medication and/or traditional/herbal ingredients which, in the opinion of the investigator, may affect study outcomes. For example, drugs or supplements containing metal ions known to impart staining to the enamel.
* Participants who have the following dental exclusions: a) Received a dental prophylaxis within 8 weeks of screening. b) Gross periodontal disease, treatment of periodontal disease (including surgery) within 12 months of screening, scaling or root planning within 3 months of screening. c) Dental conditions / disease requiring immediate treatment. d) Used any professionally dispensed or over the counter bleaching/ whitening products (excluding daily use whitening dentifrices) within the past 3 months.
* Participants who have the following specific dental exclusions for assessment teeth: a) Any tooth which, in the opinion of the investigator, appears to be non-vital based on changes in the intrinsic colour. b) Tooth with evidence of current or recent caries, or reported treatment of decay in 12 months of screening. c) Tooth with exposed dentine which, in the opinion of the investigator, could impact grading of extrinsic dental stain; tooth with deep, defective or facial restorations; tooth used as an abutment for fixed or removable partial dentures; tooth with full crown or veneer, orthodontic bands or cracked enamel. d) Tooth with surface irregularities, discoloration due to trauma, tetracycline stain, restorations, or hypo or hyperplasic areas which, in the opinion of the investigator, would prevent consistent grading of extrinsic dental stain. e) High levels of calculus deposits which might interfere with plaque assessments at the discretion of the investigator. f) Presence of orthodontic bands or appliances, extensive crowns, partial dentures, or fixed retainers.
* Any participant who, in the judgment of the investigator, should not participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2017-12-02 (Actual); Study Completion 2017-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one center in USA
Pre-assignment Details: A total of 137 participates were screened, out of which 123 participants were enrolled and randomized in the study. 14 participants were not randomized as 11 participants did not meet study criteria, 2 participants withdrew by consent and 1 participant was lost to follow-up.
Groups:
- Test Product 1: Participants were instructed to apply experimental dentifrice containing 5% potassium nitrate (KNO3) / 0.2542% sodium fluoride (NaF) dentifrice with 0.5% spherical silica.
- Test Product 2: Participants were instructed to apply experimental dentifrice containing 5% KNO3 / 0.2542% NaF dentifrice with 1% spherical silica and 5% sodium tripolyphosphate (STP).
- Reference Product 1: Participants were instructed to apply marketed dentifrice containing 5% KNO3 / 0.2542% NaF dentifrice with 6% abrasive silica.
- Reference Product 2: Participants were instructed to apply marketed dentifrice containing 5% KNO3 / 0.2543% NaF dentifrice with 16% abrasive silica and 5% STP.
Period: Overall Study
Arm/Group | Test Product 1 | Test Product 2 | Reference Product 1 | Reference Product 2
Started | 31 | 31 | 30 | 31
Completed | 31 | 31 | 30 | 30
Not Completed | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population (N=123) comprised of all participants who were randomized and received at least one dose of study treatment during the study. This population was based on the treatment the participant actually received.
Groups:
- Test Product 1: Participants were instructed to apply experimental dentifrice containing 5% KNO3) / 0.2542% NaF dentifrice with 0.5% spherical silica.
- Test Product 2: Participants were instructed to apply experimental dentifrice containing 5% KNO3 / 0.2542% NaF dentifrice with 1% spherical silica and 5% STP.
- Total: Total of all reporting groups
Arm/Group | Test Product 1 | Test Product 2 | Reference Product 1 | Reference Product 2 | Total
Number analyzed (Participants) | 31 | 31 | 30 | 31 | 123
Age, Customized [Mean (Standard Deviation); unit: Years] | 45.5 (11.32) | 46.2 (12.42) | 41.3 (11.25) | 42.9 (10.57) | 44.0 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 23 | 19 | 23 | 91
  Male | 5 | 8 | 11 | 8 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 31 | 30 | 30 | 29 | 120
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 3 | 2 | 14
  White | 24 | 27 | 27 | 28 | 106
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Overall Macpherson Modification of the Lobene Stain Index (MLSI) at 8 Weeks.
Description: An assessment of the area and intensity of dental stain on the study teeth was performed using the MLSI to evaluate ranking order in extrinsic dental stain removal or reduction of test product 1, test product 2, reference product 1, reference product 2; after usage for 8 weeks, twice daily brushing. The intensity of stain was scored separately for the gingival and body areas of each assessable tooth on a scale of 0 to 3 (0 - no stain, 1- light stain, 2 - moderate stain, 3 - heavy stain). The area of stain was scored separately for the gingival and body areas of each assessable tooth on the following scale: 0 - no stain; 1 - stain up to 1/3 of the area affected; 2- stain between 1/3 and 2/3 of the area affected; and 3 - stain more than 2/3 of area affected. Overall MLSI was calculated by multiplying scores of intensity and area, and was thus analyzed on a scale of 0 (best score) to 9 (worst score).
Time Frame: Baseline, Week 8 post treatment administration
Population: The Intent-to-Treat (ITT) (n=123) population comprised all participants who were randomly allocated to treatment and received the study treatment at least once and provided at least 1 post-baseline (post-treatment) assessment of efficacy. This population was based on the randomized treatment to which the participant was allocated.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Groups:
- Test Product 1: Participants were instructed to apply experimental dentifrice containing 5% KNO3 / 0.2542% NaF dentifrice with 0.5% spherical silica.
Arm/Group | Test Product 1 | Test Product 2 | Reference Product 1 | Reference Product 2
Number analyzed (Participants) | 31 | 31 | 30 | 31
Score on a scale | -0.32 (0.090) | -0.47 (0.090) | -0.38 (0.091) | -0.40 (0.090)
Statistical Analysis 1: Comparison: Test Product 1 vs Reference Product 1; Test type: Other; p = 0.6499, ANCOVA; From ANCOVA with treatment as fixed effect and baseline overall MLSI score as a covariate; Difference of Least Mean Square = 0.06, 95% CI 2-sided [-0.19 to 0.31], Standard Error of Mean 0.128; The reason for entering same analysis for primary and secondary is because statistical analysis was not done separately for primary outcome measure. The decision was clinical decision at the time of protocol design.There was no comparisons for the primary objective as the main objective was to look at the rank order of the treatments in level of stain reduction after 8 weeks of treatment. This was achieved via the adjusted means and confidence intervals for the means along with plots of MLSI over time. The hypothesis was that the test products would reduce stain to a greater extent than the reference products. Two comparisons of interest were done under secondary and exploratory objectives
Statistical Analysis 2: Comparison: Test Product 2 vs Reference Product 2; Test type: Other; p = 0.5680, ANCOVA; From ANCOVA with treatment as fixed effect and baseline overall MLSI score as a covariate; Difference of Least Square mean = -0.07, 95% CI 2-sided [-0.33 to 0.18], Standard Error of Mean 0.128 — -0.33 to 0.18

2. Secondary Outcome: Difference of Least Square Mean of Change From Baseline in Overall MLSI After 8 Weeks (Test Product 1 Versus vs. Reference Product 1)
Description: An assessment of the area and intensity of dental stain on the study teeth will be performed using the MLSI after usage test product 1 and reference product 1 for 8 weeks, twice daily brushing. The intensity of stain was scored separately for the gingival and body areas of each assessable tooth on a scale of 0 to 3 (0 - no stain, 1- light stain, 2 - moderate stain, 3 - heavy stain). The area of stain was scored separately for the gingival and body areas of each assessable tooth on the following scale: 0 - no stain; 1 - stain up to 1/3 of the area affected; 2- stain between 1/3 and 2/3 of the area affected; and 3 - stain more than 2/3 of area affected. Overall MLSI will be calculated by multiplying scores of intensity and area, and will be thus analyzed on a scale of 0 (best score) to 9 (worst score).
Time Frame: Baseline, Week 8 post treatment administration
Population: The ITT population comprised all participants who were randomly allocated to treatment and received the study treatment at least once and provided at least 1 post-baseline (post-treatment) assessment of efficacy. This population was based on the randomized treatment to which the participant was allocated.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Groups:
- Test Product 1 vs Reference Product 1: Participants were instructed to apply experimental dentifrice containing 5% KNO3 / 0.2542% NaF dentifrice with 0.5% spherical silica and marketed dentifrice containing 5% KNO3 / 0.2542% NaF dentifrice with 6% abrasive silica.
Arm/Group | Test Product 1 vs Reference Product 1
Number analyzed (Participants) | 61
Score on a scale | 0.06 (0.128)
Statistical Analysis 1: Comparison: Test Product 1 vs Reference Product 1; Test type: Other; p = 0.6499, ANCOVA; From ANCOVA with treatment as fixed effect and baseline overall MLSI score as a covariate; Difference of Least Square mean = 0.06, 95% CI 2-sided [-0.19 to 0.31], Standard Error of Mean 0.128 — Difference is first named treatment minus second named treatment such that a negative difference favors the first named treatment

3. Secondary Outcome: Difference of Least Square Mean of Change From Baseline in Overall MLSI After 8 Weeks (Test Product 2 Versus vs. Reference Product 2)
Description: An assessment of the area and intensity of dental stain on the study teeth will be performed using the MLSI after usage test product 2 and reference product 2 for 8 weeks, twice daily brushing. The intensity of stain was scored separately for the gingival and body areas of each assessable tooth on a scale of 0 to 3 (0 - no stain, 1- light stain, 2 - moderate stain, 3 - heavy stain). The area of stain was scored separately for the gingival and body areas of each assessable tooth on the following scale: 0 - no stain; 1 - stain up to 1/3 of the area affected; 2- stain between 1/3 and 2/3 of the area affected; and 3 - stain more than 2/3 of area affected. Overall MLSI will be calculated by multiplying scores of intensity and area, and will be thus analyzed on a scale of 0 (best score) to 9 (worst score).
Time Frame: Baseline, Week 8 post treatment administration
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Groups:
- Test Product 2 vs Reference Product 2: Participants were instructed to apply experimental dentifrice containing 5% KNO3 / 0.2542% NaF dentifrice with 1% spherical silica and 5% STP and marketed dentifrice containing 5% KNO3 / 0.2543% NaF dentifrice with 16% abrasive silica and 5% STP.
Arm/Group | Test Product 2 vs Reference Product 2
Number analyzed (Participants) | 62
Score on a scale | -0.07 (0.128)
Statistical Analysis 1: Comparison: Test Product 2 vs Reference Product 2; Test type: Other; p = 0.5680, ANCOVA; From ANCOVA with treatment as fixed effect and baseline overall MLSI score as a covariate; Difference of Least Square mean = -0.07, 95% CI 2-sided [-0.33 to 0.18], Standard Error of Mean 0.128 — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Test Product 1 | Test Product 2 | Reference Product 1 | Reference Product 2
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31 | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/31 | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 3/31 | 1/31 | 2/30 | 0/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test Product 1 (N=31) | Test Product 2 (N=31) | Reference Product 1 (N=30) | Reference Product 2 (N=31)
TRAUMATIC ULCER (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
LIP ULCERATION (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
MOUTH ULCERATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PALATAL ULCER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANGULAR CHEILITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT03267511/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT03267511/SAP_001.pdf